CLINICAL TRIAL: NCT00627432
Title: Phase 2 Randomized Study Evaluating the Efficacy of Gemcitabine With or Without Oxaliplatin in Patients With Advanced Urothelial Cancer That Cannot be Treated With Cisplatin-based Chemotherapy
Brief Title: Gemcitabine With Or Without Oxaliplatin in Treating Patients With Locally Advanced or Metastatic Bladder Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000574179; CLCC-VESUNFIT; RECF0368; SANOFI-AVENTIS-CLCC-VESUNFIT; LILLY-CLCC-VESUNFIT
Record Dates: First submitted 2008-02-29; First posted 2008-03-03 (Estimated); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Bladder Cancer
Keywords: stage III bladder cancer; stage IV bladder cancer; transitional cell carcinoma of the bladder
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Gemcitabine; Oxaliplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gemcitabine, (Active Comparator): •Arm I: Patients receive gemcitabine hydrochloride IV over 120 minutes on days 1, 8, and 15.
  Interventions: Drug: gemcitabine hydrochloride
- Gemcitabine, Oxaliplatine (Experimental): •Arm II: Patients receive gemcitabine IV over 100 minutes on days 1 and 15 and oxaliplatin IV over 120 minutes on days 2 and 16.
  Interventions: Drug: gemcitabine hydrochloride; Drug: oxaliplatin

INTERVENTIONS:
Drug: gemcitabine hydrochloride
Drug: oxaliplatin
  Arms: Gemcitabine, Oxaliplatine

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as gemcitabine and oxaliplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells.

PURPOSE: This randomized phase II trial is studying how well giving gemcitabine together with oxaliplatin works compared to gemcitabine alone in treating patients with locally advanced or metastatic bladder cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the objective response rate in patients with advanced urothelial cancer treated with gemcitabine hydrochloride with vs without oxaliplatin.

Secondary

* Determine the tolerance of these regimens in these patients.
* Determine the overall survival and progression-free survival of patients treated with these regimens.
* Determine the quality of life of patients treated with these regimens.
* Determine the duration of response in patients treated with these regimens.

OUTLINE: This is a multicenter study. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive gemcitabine hydrochloride IV over 120 minutes on days 1, 8, and 15.
* Arm II: Patients receive gemcitabine IV over 100 minutes on days 1 and 15 and oxaliplatin IV over 120 minutes on days 2 and 16.

Treatment in both arms repeats every 4 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 3 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed urothelial carcinoma, or transitional cell carcinoma of the bladder or upper urinary tract

  * Locally advanced disease (T4b) or metastatic disease (N2, N3, or M1)
* Unable to receive cisplatin-based chemotherapy due to creatinine clearance 30-60 mL/min or performance status 2
* At least 1 unidimensionally measurable lesion according to RECIST criteria
* No nonmeasurable lesions only, including any of the following:

  * Ascites
  * Pleural or pericardial effusion
  * Bone metastases
  * Lymphangitis
* No symptomatic cerebral metastases unless they have been stabilized

PATIENT CHARACTERISTICS:

* See Disease Characteristics
* Performance status 0-2
* ANC ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Alkaline phosphatase ≤ 2 times normal (unless bone metastases are present)
* Transaminases ≤ 2 times normal (5 times normal if hepatic metastases present)
* Bilirubin ≤ 1.5 times normal
* Not pregnant or nursing
* Fertile patients must use effective contraception during and for at least 6 months after completion of treatment
* No prior malignancy within the past 5 years except carcinoma in situ of the cervix or basal cell skin cancer
* No peripheral neuropathy ≥ grade 2
* No uncontrolled infection
* No other medical conditions that could interfere with evaluating tolerability, including any of the following:

  * Congestive heart failure
  * Angina pectoris that cannot be stabilized with medication
  * Myocardial infarction within the past 12 months
  * Serious thromboembolic disease
* No psychologic, social, or geographic reason that would make follow-up impossible

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior chemotherapy for advanced disease
* More than 4 weeks since prior radiotherapy to a target measurable lesion

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2004-07; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Objective response rate | From baseline to the end of treatment, up to 6 months

SECONDARY OUTCOMES:
Adverse events according to Common Terminology Criteria for Adverse Events (CTCAE) | From baseline to the end of treatment, up to 6 months
Overall survival | From baseline to the end of treatment, up to 6 months
Progression-free survival | From baseline to the end of treatment, up to 6 months
Quality of life as assessed by QLQ-C30 and QLQ-LC13 | From baseline to the end of treatment, up to 6 months
Duration of response | From baseline to the end of treatment, up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Damien Pouessel, MD, Study Chair — Institut du Cancer de Montpellier - Val d'Aurelle
Locations (1):
- Centre Regional de Lutte Contre le Cancer - Centre Val d'Aurelle, Montpellier, France